CLINICAL TRIAL: NCT04742127
Title: Failure of a Single Surgical Debridement in Septic Arthritis of the Native Hip: a Retrospective Study
Brief Title: Failure of a Single Surgical Debridement in Septic Arthritis of the Native Hip
Status: Active, not recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S64930
Record Dates: First submitted 2021-01-29; First posted 2021-02-05 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Septic Arthritis of the Native Hip; Failure of Initial Debridement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with septic arthritis of the native hip
  Interventions: Diagnostic Test: Single surgical debridement

INTERVENTIONS:
Diagnostic Test: Single surgical debridement — To describe the clinical factors associated with failure of a single surgical debridement in patients with septic arthritis of the native hip.

SUMMARY:
Septic arthritis of the native hip poses significant diagnostic and therapeutic challenges as it is considered an orthopedic emergency requiring urgent surgery. Inadequate or delayed treatment is disastrous, resulting in irreversible destruction of the joint. Initial treatment usually comprises of arthroscopic or open debridement. According to literature 25-38% of first debridement fail, requiring a second or third intervention or even a staged procedure with femoral head resection and a temporary antibiotic-loaded cement spacer.

Understanding who will succeed and who will fail after a single surgical debridement of a septic hip joint could improve shared decision-making and could help decide which patient would benefit from resection arthroplasty straight away.

In order to gain more insight in clinical factors associated with failure of a single surgical debridement in septic arthritis of the native hip, a retrospective cohort study will be conducted. There are no detailed guidelines for the treatment of septic arthritis of the native hip. Therefore, treatment today is similar to treatment 10 years ago (i.e. the treating surgeon does what he thinks is best for the patient). This lack of a structured approach is the reason for this retrospective study and we aim to come up with principles to guide treatment of future patients.

DETAILED DESCRIPTION:
Septic arthritis of the native hip poses significant diagnostic and therapeutic challenges as it is considered an orthopedic emergency requiring urgent surgery. Early diagnosis remains difficult as the golden standard is based on microbiological confirmation of bacteria in synovial fluid or solid tissue biopsies, which can take up to a minimum of 3-5 days or longer. Inadequate or delayed treatment is disastrous, resulting in irreversible destruction of the joint. Initial treatment usually comprises of arthroscopic or open debridement. In comparison to septic arthritis of the knee, patients are more often less fit and the joint is less accessible for arthroscopic intervention. Initial surgical debridement should be performed within 24 hours of occurrence. According to literature 25-38% of first debridement fail, requiring a second or third intervention or even a staged procedure with femoral head resection and a temporary antibiotic-loaded cement spacer.

Understanding who will succeed and who will fail after a single surgical debridement of a septic hip joint could improve shared decision-making and could help decide which patient would benefit from resection arthroplasty straight away. Factors such as a history of inflammatory arthritis, diabetes, a synovial-fluid nucleated cell count of > 85.0 x 10^9 cells/L, S. aureus, delay to surgery and positive cultures of drain fluid were associated with failure of initial debridement, but have not been validated. Considering the increased use of MRI and nuclear imaging in the work-up of these patients, there might be additional useful risk factors, such as extra-articular manifestation of the infection, AVN of the femoral head, severe degeneration of the joint, multi-joint involvement, SUV-max values on FDG-PET-CT and so on.

Most literature surrounding this subject is limited to case reports and case series with small sample sizes. Due to the sizable amounts of tertiary references, a large population of transplant patients treated at the institution UZ Leuven Gasthuisberg, and the own experience of the investigators, the investigators are convinced that the population size at is substantially larger.

In order to gain more insight in clinical factors associated with failure of a single surgical debridement in septic arthritis of the native hip, a retrospective cohort study will be conducted. There are no detailed guidelines for the treatment of septic arthritis of the native hip. Therefore, treatment today is similar to treatment 10 years ago (i.e. the treating surgeon does what he thinks is best for the patient). This lack of a structured approach is the reason for this retrospective study and we aim to come up with principles to guide treatment of future patients.

ELIGIBILITY:
Inclusion Criteria:

* All microbiology reports for cases of septic arthritis of the native hip joint concerning synovial fluid or solid tissue cultures obtained from arthrocentesis/debridement of the hip, collected from January 1st 2010 to January 1st 2020
* Patients are at least 18 years of age
* Cases with positive cultures in patients of which the initial diagnosis, treatment and follow-up was conducted at UZ Leuven Gasthuisberg

Exclusion Criteria:

- History of arthroplasty of the hip in the affected joint

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with septic arthritis of the native hip treated at UZ Leuven in the last decade
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical factors associated with failure of a single surgical debridement | Through study completion, an average of 1 year
  A retrospective data registry containing clinical data of patients with septic arthritis of the native hip will be constructed. This data registry will contain a sizable amount of clinico-pathological features collected from the electronic patient registry. Subsequently, a retrospective cohort study will be conducted in order to establish associations between certain clinical factors and the likelihood of failure of the initial surgical debridement.

SECONDARY OUTCOMES:
Population of patients who would benefit from a staged procedure | Through study completion, an average of 1 year
  A proportion analysis will be conducted in order to find typical characteristics present in patients with septic arthritis of the native hip. These characteristics will be used to find and describe a subpopulation of patients who would benefit from a staged procedure with femoral head resection and a temporary antibiotic-loaded cement spacer followed by total hip arthroplasty straight away, instead of initial debridement of the native hip.
Prevalence of failure of initial debridement | Through study completion, an average of 1 year
  The prevalence of failure of initial debridement will be described using the retrospective dataset.
Prevalence of staged procedure | Through study completion, an average of 1 year
  The prevalence of patients needing a staged procedure will be described using the retrospective dataset.
Mortality | Through study completion, an average of 1 year
  The mortality rate after treatment will be described using the retrospective dataset.
Recurrence | Through study completion, an average of 1 year
  The recurrence rate after treatment will be described using the retrospective dataset.
Risk factors for failure of a single surgical debridement | Through study completion, an average of 1 year
  Risk factors for failure of a single surgical debridement will be identified using the predictive model developed by Hunter et al. This predictive model is a prognostic probability algorithm to predict failure of a single surgical debridement.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided